CLINICAL TRIAL: NCT01012752
Title: A Multicenter, Double-Blind, Placebo-Controlled Study With a Modified Allergen Extract for Specific Immunotherapy in Patients With Seasonal Allergic Rhinitis/Rhinoconjunctivitis
Brief Title: A Multicenter Study to Evaluate Safety and Efficacy of Specific Immunotherapy With Modified Allergen Extracts
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Roxall Medizin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBC-2009-003B
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Allergic Rhinitis; Allergic Conjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- modified allergen extract (Active Comparator)
  Interventions: Biological: modified allergen extract
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: modified allergen extract — subcutaneous injections
  Arms: modified allergen extract
Biological: Placebo — subcutaneous injections
  Arms: Placebo

SUMMARY:
This trial is performed to evaluate the safety and clinical efficacy of subcutaneous specific immunotherapy in patients suffering from seasonal allergic rhinitis/rhinoconjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Positive history of allergen specific allergic rhinitis/rhinoconjunctivitis
* Positive screening skin prick test (wheal diameter > 3 mm)
* Compliance and ability of the patient to complete a Diary Card for self-evaluating of the symptoms and antisymptomatic medication
* Signed and dated patient´s Informed Consent,

Exclusion Criteria:

* Previous immunotherapy within the last 3 years,
* Simultaneous participation in other clinical trials,
* Other reasons contra-indicating an inclusion into the trial according to the investigator´s estimation (e.g. poor compliance),
* Auto-immune disorders,
* Severe chronic inflammatory diseases,
* Malignancy,
* Alcohol abuse,
* Existing or intended pregnancy, lactation and/or lack of adequate contraceptive protection,
* Treatment with beta-blockers (incl. local application) and/or other contra-indicated drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Symptom and medication score | 1 year

SECONDARY OUTCOMES:
Safety of the treatment | 1 year
Documentation of adverse events | 1 year
Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | 1 year
Clinical global improvement | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hamburg, Germany